CLINICAL TRIAL: NCT01747720
Title: A Randomized Double-blind Placebo-controlled Trial of the Effect of Vitamin D Supplementation on Breast Density in Premenopausal Women
Brief Title: Vitamin D and Mammographic Breast Density
Acronym: EVIDENSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Quebec Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DR-002-1373
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; mammographic breast density; vitamin D; prevention; randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D3 (cholecalciferol) 1000 IU (Experimental): Oral vitamin D3 (cholecalciferol) supplementation, 1000 IU daily, for 12 months
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 (cholecalciferol) 2000 IU (Experimental): Oral vitamin D3 (cholecalciferol) supplementation, 2000 IU daily, for 12 months
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 (cholecalciferol) 3000 IU (Experimental): Oral vitamin D3 (cholecalciferol) supplementation, 3000 IU daily, for 12 months
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): daily, for 12 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Given orally
  Other Names: Cholecalciferol
  Arms: Vitamin D3 (cholecalciferol) 1000 IU; Vitamin D3 (cholecalciferol) 2000 IU; Vitamin D3 (cholecalciferol) 3000 IU
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
There is some evidence that vitamin D could be used to reduce breast cancer risk. Randomized controlled trials would provide definitive evidence about this effect. However, trials with breast cancer as outcome are expensive and time-consuming. Use of surrogate outcomes has been advocated to accelerate progress in the identification of interventions that could prevent breast cancer. Mammographic breast density is one of the strongest breast cancer risk indicators and is already used as a surrogate outcome in several breast cancer prevention trials. The aim of this double-blind randomized controlled trial is to determine whether daily oral supplementation with vitamin D3 (1,000, 2,000 or 3,000 IU) over a period of 1 year reduces breast density in premenopausal women compared to placebo. A total of 376 women (94 per arm) who live in Quebec City will be recruited. Showing that vitamin D reduces breast density would provide strong support for the idea that vitamin D can be a safe and inexpensive approach for the prevention of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES

Primary:

- to determine whether adding oral supplementation with vitamin D3 (cholecalciferol) at doses of 1,000, 2,000 and 3,000 IU/d to baseline total vitamin D intake over a period of 12 months reduces mammographic breast density among premenopausal women at moderate to high risk of breast cancer who reside in the Quebec City area, Canada.

Secondary:

* to assess the net increase in 25(OH)D levels resulting from this vitamin D3 supplementation;
* to document the compliance with, and safety of, supplementation with tested doses of vitamin D3 over one year.

OUTLINE This study is a double-blind, placebo-controlled, randomized trial among premenopausal women who live in the Quebec City area and have ≥ 20% breast density at baseline.

The intervention consists of the addition, over baseline total vitamin D intake from food and supplements, of three different doses of vitamin D3 (1000, 2000 or 3000 IU/day) for a period of 12 months. There are four arms in the trial:

* Arm 1: 1,000 IU vitamin D3/d (1 tablet vitamin D 1000 IU + 2 tablets placebo);
* Arm 2: 2,000 IU vitamin D3/d (2 tablets vitamin D 1000 IU + 1 tablet placebo);
* Arm 3: 3,000 IU vitamin D3/d (3 tablets vitamin D 1000 IU);
* Arm 4: placebo (3 tablets placebo/d).

Vitamin D tablets (1000 IU tablets) and the placebo tablets are undistinguishable in size, shape, color and taste, and are manufactured by the same company.

ELIGIBILITY:
Inclusion Criteria:

* be premenopausal at baseline;
* have breast density of at least 20% at baseline;
* have normal baseline serum calcium (2,12-2,60 mmol/L) and serum creatinine (45-85 μmol/L);
* agree to have her mammogram at 12 months of follow-up at the same mammography clinic (same site) as the one where the mammogram at recruitment was done.

Exclusion Criteria:

* taking > 400 IU/day of supplemental vitamin D and refusing to reduce (≤ 400 IU/day) or cease such intake;
* taking > 600 mg/day of supplemental calcium and refusing to reduce (≤ 600 mg/day) or cease such intake;
* have contra-indications for use of vitamin D supplementation (hypersensitivity to vitamin D or its analogues; a history of renal calculi or hypercalcemia, hypervitaminosis D);
* taking medication suspected to interact with vitamin D: frequent use of antacids containing magnesium or aluminium; regular use of anticonvulsants (phenytoin, phenobarbital), digoxin, cholestyramine, colestipol, orlistat, mineral oil;
* have a personal history of breast cancer;
* have a personal history of cancer other than non-melanoma skin cancer within 5 last years;
* have had breast reduction or augmentation including breast implantation (or planning to undergo such surgery during the trial);
* be pregnant or planning a pregnancy in the next year.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 405 (Actual)
Dates: Start 2012-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Mammographic breast density | 12 months
  Difference in breast density between baseline and at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Brisson, M.D., Sc.D., Principal Investigator — Centre de recherche du CHU de Québec, et Faculté de médecine de l'Université Laval
Locations (1):
- Centre de recherche du CHU de Québec, Hôpital du Saint-Sacrement, Québec, Canada

IPD SHARING:
Plan to Share IPD: No
We will not share IPD. Results of the study are published in Cancer Epidemiology, Biomarkers and Prevention.